CLINICAL TRIAL: NCT03381014
Title: Added Benefit of Speckle Tracking Echo to Molecular Expression of High Sensitive Troponin I and Cardiac Ryanodine Receptor in Early Detection of Cardiomyopathy in Patients Receiving Anthracycline Chemotherapy
Brief Title: Early Detection of Cardiomyopathy by Speckle Echo, High Sensitive Troponin and Cardiac Ryanodine Receptors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Mahmoud Morsy, doctor, Assiut University
Other Study IDs: speckle echo in cardiomyopathy
Record Dates: First submitted 2017-12-12; First posted 2017-12-21 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Chemotherapy Effect
MeSH Terms: interventions — Anthracyclines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: Chemotherapy, Cancer, Anthracyclines — follow up cardio-toxicity .... by speckle tracking echo and cardiac troponin
  Other Names: speckle tracking Echo

SUMMARY:
Early detection of cardiomyopathy in patients receiving Anthracycline chemotherapy and determine if speckle tracking echo and Troponin gene will add benefit for early detection of cardiomyopathy.

Improve economic impact of oncologic patients from whom high sensitive troponin negative and normal speckle tracking patients can be safely excluded from long-term cardiac monitoring programs.

To correlate between the molecular gene expression of troponin genes and ryanodine receptor in cardiomyopathy

DETAILED DESCRIPTION:
Anthracycline chemotherapy has saved the lives of many cancer victims during the 50 years after their discovery.These patients are prone to higher risk of cardiovascular death than the risk of tumor recurrence, particularly in childhood cancer survivors in whom the cardiac mortality rate is seven fold higher.

Cardiac toxicity remains an important side effect of anticancer therapies, leading to increased mortality due to mainly heart failure, but also arrhythmias, hypertension, thromboembolism.

The time from early development of cardiac dysfunction to the modification or end of chemotherapy and beginning of heart failure therapy, is an important determinant of the extent of recovery.

The Cardiotoxicity of anthracyclines may be acute, early or late. A recent study involving 2625 patients (mean follow-up 5 years); showed a 9% overall incidence of Cardiotoxicity after anthracycline treatment, 98% of cases occurred within the first year and were asymptomatic.

Cardiotoxicity has been defined using various classifications. Recent guidelines suggest that Cancer therapeutics-related cardiac dysfunction (CTRCD) is defined as a decrease in the LVEF (by echocardiography) of >10 percentage points to a value below the lower limit of normal.

Echocardiography should be repeated before every next administration of anthracycline, after 3, 6, and 12 months from the end of therapy with anthracycline but...Not all patients treated with chemotherapy require such frequently repeated LVEF monitoring as suggested by the guidelines because of the negative impact on patient management and cost-effectiveness ratio for the national health system.

Speckle-tracking echocardiography is a noninvasive ultrasound imaging technique that allows for early an objective and quantitative evaluation of global and regional myocardial function.

New elevation of serum troponin detected with high sensitivity Troponin assays in patients receiving anthracyclines also predicts subsequent LV dysfunction.

Ryanodine receptors (RyRs) are a class of intracellular calcium channels in various forms of excitable tissues like muscles and neurons.

In heart failure the RyR2 channels become abnormally active or "leaky" and are unable to remain closed during diastole. This leads to an increase in spontaneous Ca+2 spark frequency and dysregulated Ca+2 handling within the cardiomyocyte, resulting in decreased systolic contraction and irregular contractile activity.

ELIGIBILITY:
Inclusion Criteria:

* all Newly diagnosed cancer patients with who will receive Anthracycline based regimen chemotherapy

Exclusion Criteria:

* Insufficient ultrasound image quality, defined as more than three LV segments being suboptimally visualized by conventional echocardiography.
* Valvular heart disease
* Hypertensive heart disease
* Cardiomyopathy
* Chronic renal failure
* Chronic obstructive air way disease (COPD)

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Cancer patient between the age of 30-50yr who will receive chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
early detection of cardiomyopathy | about one year
  using speckle tracking echo to early diagnosis of cardiomyopathy
identify patients whose at risk to develop cardiomyopathy | about one year
  Using the high sensitive troponin with quantitative measurements as biomarker.

SECONDARY OUTCOMES:
molecular gene expression of troponin genes and ryanodine receptor in cardiomyopathy | same time frame ... about one year
  quantitative correlation between the troponin genes and ryanodine receptor in early cardiomyopathy

CONTACTS AND LOCATIONS:
Overall Officials: yehia T kishk, MD, Study Chair — cardiology department; Mohamed K Koriem, MD, Principal Investigator — cardiology department; Naglaa K Idriss, MD, Principal Investigator — biochemistry department

REFERENCES:
- [Result] Henning RJ, Harbison RD. Cardio-oncology: cardiovascular complications of cancer therapy. Future Cardiol. 2017 Jul;13(4):379-396. doi: 10.2217/fca-2016-0081. Epub 2017 Jun 29. PMID 28660778
- [Result] Curigliano G, Cardinale D, Dent S, Criscitiello C, Aseyev O, Lenihan D, Cipolla CM. Cardiotoxicity of anticancer treatments: Epidemiology, detection, and management. CA Cancer J Clin. 2016 Jul;66(4):309-25. doi: 10.3322/caac.21341. Epub 2016 Feb 26. PMID 26919165
- See also: Cancer Chemotherapy and Cardiac Arrhythmias: A Review — http://www.readcube.com/articles/10.1007/s40264-014-0258-4